CLINICAL TRIAL: NCT06260579
Title: A Home-based Exercise and Physical Activity Intervention After Kidney Transplantation: Impact of Exercise Intensity - a Multicenter Randomized Controlled Trial
Brief Title: Home-based Exercise and Physical Activity Intervention After Kidney Transplantation: Impact of Exercise Intensity
Acronym: PHOENIX-Kidney
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: University Ghent (Other)
Responsible Party: Principal Investigator, Amaryllis Van Craenenbroeck, Professor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: S-number 66153; S006722N (Other Grant/Funding Number: Research Foundation Flanders - SBO project)
Record Dates: First submitted 2024-01-25; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Physical Activity; Exercise Training; Kidney Transplantation; Physical Fitness; Cardiovascular Health; Gut Microbiome; Health-related Quality of Life; Implementation; Cost-effectiveness
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Parallel group randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are blinded to the group allocation of the patients. Due to the nature of the intervention, blinding of the patients is not possible. However, a sham training intervention is provided to the control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low intensity training (LIT) (Sham Comparator): 6 months of low-intensity flexibility and balance exercises, not followed by a formal physical activity intervention
  Interventions: Behavioral: Exercise/physical activity
- Moderate-intensity training (MIT) (Experimental): 6 months of exercise intervention (moderate intensity), followed by a co-developed physical activity intervention
  Interventions: Behavioral: Exercise/physical activity
- Moderate- and high-intensity training group (MHIT) (Experimental): 6 months of exercise intervention (moderate-intensity followed by high-intensity), followed by a co-developed physical activity intervention
  Interventions: Behavioral: Exercise/physical activity

INTERVENTIONS:
Behavioral: Exercise/physical activity — personalized exercise training and physical activity program

SUMMARY:
This multicentre two-phased RCT aims to evaluate implementation potential, cost-effectiveness, effectiveness, and the role of exercise intensity of a home-based exercise and physical activity intervention to improve de novo kidney transplant recipients' physical fitness, cardiovascular health, gut microbiome characteristics, and health-related quality of life. The first phase of this study comprehends a six-month exercise training intervention. Patients will be randomized into (i) a sham intervention consisting of low-intensity balance and stretching exercises (LIT), (ii) a moderate-intensity aerobic and strength training intervention (MIT), or (iii) a moderate- and high-intensity aerobic and strength training intervention (MHIT). The second phase of this study comprehends a physical activity maintenance intervention provided to MIT and MHIT but not LIT. A total of 147 de novo kidney transplant recipients will be recruited from two independent Belgian transplant centres i.e. UZ Leuven and UZ Ghent.

DETAILED DESCRIPTION:
Advances in the field of kidney transplantation have led to improved postoperative survival rates, but age-standardized mortality nonetheless remains two to sevenfold higher in kidney transplant recipients - with cardiovascular disease representing the leading cause of death in recipients with a functioning graft. Poor physical fitness, not completely recovering after transplantation, adds to the heightened cardiovascular risk of hypertension, diabetes, dyslipidaemia, and obesity. So does the posttransplant continuation of gut microbial dysbiosis, which recently emerged as a modulator of muscular, metabolic, and cardiovascular health. Exercise-based rehabilitation and physical activity interventions may prove pivotal in the care of kidney transplant recipients to address aforementioned outcomes.

This multicentre two-phased RCT comprehends a six-month exercise intervention at different exercise intensities, followed by an implementation strategy bundle promoting a physically active lifestyle. A total of 147 adult de novo kidney transplant recipients from two independent Belgian transplant centres will be randomly allocated to either 6 months of home-based exercise training consisting of muscle flexibility and postural stability exercises (low intensity training, LIT, n=49), moderate-intensity aerobic and strength training (moderate intensity training, MIT, n=49), or moderate- and high-intensity aerobic and strength training (moderate- and high-intensity training, MHIT, n=49). MIT will participate in moderate-intensity aerobic training on a stationary bicycle thrice a week and moderate-intensity strength training sessions twice a week. During the initial three months of the exercise intervention MHIT will participate in the same training program as MIT. In the final three months of the training intervention, MHIT will participate in high-intensity aerobic training on a stationary bicycle thrice a week and moderate-intensity strength training twice a week.

Following the six-month exercise training intervention, MIT and MHIT, but not LIT, will receive an individualized activity intervention aiming for long-term physical activity maintenance; using motivational interviewing techniques, co-creation of an action plan adapted to the patients' preferences, goal-setting, gradually decreasing follow-up prompts over time, and self-monitoring of physical activity behaviour. The training and physical activity interventions are initiated 3 and 9 months after transplantation, respectively. Study participants will be followed-up till 2 years after transplantation.

The investigators hypothesize that the study intervention will improve the primary outcome cardiorespiratory fitness, assessed as peak oxygen uptake, at 9 months posttransplant. Secondary outcomes include muscle fitness, motor fitness, body composition, cardiovascular health, gut microbiome characteristics, health-related quality of life, safety, cost-effectiveness, and implementation outcomes at six, nine, 12 and 24 months posttransplant. The role of training intensity and the role of baseline gut microbiome characteristics as predictor of individuals' training response will be explored.

ELIGIBILITY:
Inclusion Criteria:

De novo adult KTRs

Exclusion Criteria:

* Underlying heart disease, defined as aberrant CPET, unstable angina, non-revascularized lesions or life-threatening arrhythmias
* Uncontrolled hypertension
* Uncontrolled diabetes, defined as HbA1c ≥ 9%
* Musculoskeletal disorders not allowing physical training on a cycle ergometer, or any other medical reasons by the physician considered to be a contraindication for moderate or high-intensity physical exercise
* Multi-organ transplantation
* Ongoing treatment for malignancies
* Unable to understand Dutch
* No access to smartphone and/or computer with internet access
* Severe pulmonary disease defined as either forced vital capacity (FVC) <50%, one-second value (FEV1) <50%, or a diffusing capacity for carbon monoxide (DLCO) <40% that excludes all serious underlying respiratory disease (pulmonary fibrosis, COPD GOLD II-IV, PAH).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Changes in peak oxygen consumption (VO2peak) | 6, 12 and 24 months follow-up
  Assessed by a maximal cardiopulmonary exercise test

SECONDARY OUTCOMES:
Health-related physical fitness | 3, 6, 9, and 24 months after kidney transplantation
  6 minute walking test

CONTACTS AND LOCATIONS:
Overall Officials: Amaryllis Van Craenenbroeck, MD, PhD, Principal Investigator — KU Leuven; Patrick Calders, PhD, Principal Investigator — University Ghent
Locations (2):
- Belgium (2):
  - UZ Ghent, Ghent
  - UZ Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Smet S, Vandecruys M, De Beir J, Leunis S, Wyngaert KV, Renier M, de Loor H, Goetschalckx K, Naesens M, De Smedt D, Verbeke F, Stalmans I, Fieuws S, Glorieux G, Van Eijgen J, Van Criekinge H, Raes J, De Geest S, Van Biesen W, Kuypers D, Nagler E, Calders P, Monbaliu D, Cornelissen V, Van Craenenbroeck AH. Home-based exercise and physical activity intervention after kidney transplantation: impact of exercise intensity (PHOENIX-Kidney). Protocol for a multicentre randomized controlled trial. Clin Kidney J. 2025 Apr 24;18(11):sfaf114. doi: 10.1093/ckj/sfaf114. eCollection 2025 Nov. PMID 41215780